CLINICAL TRIAL: NCT07271212
Title: Evaluation of the Scalp Skin Care Effects of Premium Revitalizing Elixir
Brief Title: Scalp Care Efficacy Evaluation for Premium Revitalizing Elixir
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hungkuang University (Other)
Collaborators: Schweitzer Biotech Company (Unknown)
Responsible Party: Principal Investigator, Tsong-Min Chang, Vice President, Hungkuang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-090-A
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Scalp Health; Hair Condition; Hair Loss; Alopecia; Sebum Production; Hair Health; Hair Thinning
Keywords: Scalp care; Hair loss; Alopecia; Skin texture; Sebum measurement; Hair thinning; Scalp condition; Extracellular vesicles; Growth factors; Centella asiatica; Ginger; Cosmetics; hair density; Product formulation
MeSH Terms: conditions — Alopecia | interventions — Insulin-Like Growth Factor I; Centella asiatica extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1: Placebo control (Placebo Comparator): Base formula without caffeine and panthenol
  Interventions: Other: Placebo control
- Group 2: Base formula only (Experimental): Base formula consisting of active ingredients 0.1% caffeine and panthenol (vitamin B5).
  Interventions: Other: Base formula only
- Group 3: Base formula plus IGF-1 & FGF-7. (Experimental): Base formula plus insulin growth factor 1 (IGF-1) and fibroblast growth factor-7 (FGF-7)
  Interventions: Other: Base formula plus IGF-1 and FGF-7
- Group 4: Base formula plus Centella asiatica and ginger extracellular vesicles (Experimental): Base formula plus Centella asiatica and ginger (Zingiber officinale) extracellular vesicles
  Interventions: Other: Base formula plus Centella asiatica and ginger extracellular vesicles
- Group 5: Base formula plus Centella asiatica and ginger extracellular vesicles, IGF-1 & FGF-7. (Experimental): Base formula plus Centella asiatica and ginger (Zingiber officinale) extracellular vesicles, insulin growth factor-1 (IGF-1) and fibroblast growth factor-7 (FGF-7).
  Interventions: Other: Base formula plus Centella asiatica and ginger extracellular vesicles, IGF-1 & FGF-7

INTERVENTIONS:
Other: Placebo control — Placebo control (base formula without caffeine and panthenol). Applied 1mL evenly to the scalp once daily after hair wash for 56 consecutive days.
  Arms: Group 1: Placebo control
Other: Base formula only — Base formula consisting of active ingredients 0.1% caffeine and panthenol. Applied 1mL evenly to the scalp once daily after hair wash for 56 consecutive days.
  Arms: Group 2: Base formula only
Other: Base formula plus IGF-1 and FGF-7 — Base formula plus insulin growth factor 1 (IGF-1) and fibroblast growth factor-7 (FGF-7). Applied 1mL evenly to the scalp once daily after hair wash for 56 consecutive days.
  Arms: Group 3: Base formula plus IGF-1 & FGF-7.
Other: Base formula plus Centella asiatica and ginger extracellular vesicles — Base formula plus Centella asiatica and ginger extracellular vesicles. Applied 1mL evenly to the scalp once daily after hair wash for 56 consecutive days.
  Arms: Group 4: Base formula plus Centella asiatica and ginger extracellular vesicles
Other: Base formula plus Centella asiatica and ginger extracellular vesicles, IGF-1 & FGF-7 — Base formula plus Centella asiatica and ginger extracellular vesicles, insulin growth factor-1 (IGF-1) and fibroblast growth factor-7 (FGF-7). Applied 1mL evenly to the scalp once daily after hair wash for 56 consecutive days.
  Arms: Group 5: Base formula plus Centella asiatica and ginger extracellular vesicles, IGF-1 & FGF-7.

SUMMARY:
The study aims to evaluate the efficacy of the Premium Revitalizing Elixir on human scalp skin. A total of 60 healthy adults, aged 18 to 60 with alopecia, baldness, or self-identified with symptoms of hair thinning will be recruited and randomly assigned into five groups receiving different formulations. Participants will use the product once daily for 56 days, and their scalp conditions will be assessed through skin texture tests at multiple time points. Key parameters such as sebum content, overall hair loss, hair density, scalp condition, and hair length will be measured. A self-assessment and assessment by a hair specialist on hair and scalp condition will also be provided at the end of the study (Day 56).

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blinded, and placebo-controlled study to investigate the effects of Premium Scalp Revitalizing Essence on changes in the skin texture of human scalp skin.

This study aims to enroll 60 healthy adults aged from 18 to 60 with alopecia, baldness, or self-identified with symptoms of hair thinning.

Inclusion criteria include healthy adults defined as individuals without chronic diseases, significant illnesses (including cancer, post-stroke disorders, paralysis, acute myocardial infarction, coronary artery bypass surgery, end-stage renal disease, and major organ transplant or hematopoietic stem cell transplant), or allergic constitutions, and who are not currently taking any medication or using any scalp care products.

Exclusion criteria include individuals who are pregnant or breastfeeding, as well as males or females with chronic diseases, significant illnesses, or allergic constitutions, currently using scalp care products, students or employees affiliated with the principal investigator, individuals with scalp wounds, those who have participated in cosmetic product testing, and those who have undergone scalp aesthetic treatments within the past three months.

The participants will be randomly assigned into five groups, with 12 individuals in each group. Group 1 uses Placebo (Base formula without caffeine and panthenol); Group 2 uses the Base formula (Control with 0.1% caffeine and panthenol); Group 3 uses Base + IGF-1 & FGF-7; Group 4 uses Base + Centella asiatica extracellular vesicles + Ginger-derived extracellular vesicles; Group 5 uses Base + Centella asiatica extracellular vesicles + Ginger-derived extracellular vesicles + IGF-1 & FGF-7. Before using the test product, all 60 participants undergo the first scalp skin texture test. After 14 days of using the test product, a second scalp skin texture test is conducted; after 28 days of use, a third test is performed; after 42 days of use, a fourth test is conducted; and after 56 days of use, a fifth test is carried out. The scalp skin texture tests include measurements of skin (1) sebum content, (2) overall hair loss, (3) hair density, (4) scalp condition, (5) hair length, and other parameters. The Sebumeter® SM815 probe of the MPA580 device and the ScalpX Intelligent Scalp Diagnostic System will be used to measure the parameters of the study. On Day 56, the participants will be asked to fill out a self-assessment form and a hair specialist will also assess the hair and scalp condition at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of any gender from the age of 18 to 60 years (inclusive).
* Having symptoms of alopecia, baldness, or self-identified with hair thinning.
* Absence of chronic diseases, major illnesses, or allergies.
* Major illnesses include cancer, post-stroke disorders, paralysis, acute myocardial infarction, coronary artery bypass surgery, end-stage renal disease, and major organ transplant or hematopoietic stem cell transplant

Exclusion Criteria:

* Currently taking any medication or using any scalp care products
* Pregnant or breastfeeding
* Chronic diseases, significant illnesses, or allergic constitutions
* Currently using scalp care products
* Students or employees affiliated with the principal investigator,
* Individuals with scalp wounds
* Participated in cosmetic product testing
* Undergone scalp aesthetic treatments within the past three months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Sebum Content | Assessment conducted every 14 days from Day 0 to Day 56 (including Day 0 as baseline)
  Assess oil levels on the scalp at standardized scalp sites (left, right, and vertex). Measured with C+K Multi Probe Adaptor MPA580 system using the Sebumeter® SM815 probe based on the grease spot photometry method with the sebum measurement cassette tape.
Hair length | Assessment conducted every 14 days from Day 0 to Day 56 (including Day 0 as baseline)
  Hair length (cm): Measured manually with ruler at standardized scalp sites (left, right, and vertex).
Hair density | Assessment conducted every 14 days from Day 0 to Day 56 (including Day 0 as baseline)
  Hair density (number of hairs/cm-square): Assessed with the ScalpX Intelligent Scalp Diagnostic System with digital microscopy at standardized scalp sites (left, right, and vertex).
Hair thickness | Assessment conducted every 14 days from Day 0 to Day 56 (including Day 0 as baseline)
  Hair thickness (micrometers): Assessed with the ScalpX Intelligent Scalp Diagnostic System with digital microscopy at standardized scalp sites (left, right, and vertex).
Hair loss | Assessment conducted every 14 days from Day 0 to Day 56 (including Day 0)
  Hair loss: Assessed by the standardized hair combing test by counting the number of hairs shed after the participants' hair was combed over a clean surface for 60 strokes.

SECONDARY OUTCOMES:
Participant self-assessment | Day 56 (End of the study period)
  Participants will be asked to fill out an assessment form with score from 0 to 4 for each of the hair and scalp condition evaluated.
Hair specialist assessment | Day 56 (End of the study)
  A hair specialist will assess the hair and scalp condition of the participant and assign a score from 0 to 4 for each of the evaluated items as well as assign a score of Global Aesthetic Improvement Scale (GAIS) from -1 to 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Hungkuang University, Taichung, Taiwan